CLINICAL TRIAL: NCT05944406
Title: Enhancing Triage Accuracy and Streamlining Emergency Department Services: A Clinical Audit of the Manchester Triage System Implementation
Brief Title: Enhancing Triage Accuracy: A Clinical Audit of the Manchester Triage System Implementation
Status: Completed | Type: Observational
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Maham Leeza Adil, Principal Investigator, Rawalpindi Medical College
Other Study IDs: 887456
Record Dates: First submitted 2023-06-27; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Triage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Audit Cycle 1: These are the patients included in the first cycle of the clinical audit. The study collected data from a sample of 256 patients who visited the Medical Unit I of Benazir Bhutto Hospital, Rawalpindi, during the specified period. The patients were triaged by the triage nurses using the Manchester Triage System (MTS). Their age, gender, registration time, time of consultation, triage category assigned by the triage nurse, and admission decision were recorded for analysis. The accuracy of triage and waiting times were assessed for these patients.
- Audit Cycle 2: These are the patients included in the second cycle of the clinical audit, conducted after an educational intervention for the triage nurses. The study collected data from a sample of 238 patients who visited the same Medical Unit I of Benazir Bhutto Hospital, Rawalpindi. Similar to audit cycle 1, these patients were triaged using the MTS, and their demographic information, triage category, and admission decision were recorded. The study aimed to evaluate any improvements in triage accuracy and waiting times compared to audit cycle 1 after the intervention and training of the triage nurses.
  Interventions: Other: Educational training of ER Nurses

INTERVENTIONS:
Other: Educational training of ER Nurses — educational intervention was conducted from 2nd to 5th May 2023 with the triage nurses. This intervention comprised of detailed explanations of how the Triage system is accurately used to categorize the patients presenting in the ED and Triage nurses were instructed to refer non-urgent cases to either the Outpatient department or to the Casualty Medical Officer. The results of the first audit were also shared. Additionally, circulars containing instructions regarding accurate usage of MTS were distributed to all triage nurses
  Groups: Audit Cycle 2

SUMMARY:
This clinical audit focused on improving how patients are prioritized and managed in the emergency department. The audit took place in a hospital in Rawalpindi and involved two cycles of data collection. The results showed that after an educational intervention, there was an improvement in accurately triaging patients and a decrease in cases that were categorized as urgent when they were not. The audit also revealed a decrease in non-urgent cases visiting the emergency department. The findings highlight the importance of proper training, following triage guidelines, and referring non-urgent cases to other departments. The suggestions include improving the triage process and making the emergency department more efficient for better patient care.

DETAILED DESCRIPTION:
This clinical audit aimed to assess the accuracy and effectiveness of the Manchester Triage System (MTS) implementation in a hospital's emergency department. The audit took place in Medical Unit I of Benazir Bhutto Hospital, Rawalpindi, over two cycles from March to June 2023.

The hospital, affiliated with Rawalpindi Medical University, is a 750-bed tertiary care facility located in a busy city. The emergency department, equipped with approximately 91 beds, follows triage guidelines established by the hospital. The triage process involves categorizing patients based on their presenting problem and determining the time within which they should be evaluated and treated by a doctor.

To conduct the audit, certain standards were set before assessing the triage process. These included ensuring guidelines on patient categorization into triage categories, using a standard triage box in the patient record sheet, setting waiting time limits for each category, and using the discharge diagnosis of the doctor as a benchmark for triage accuracy.

The audit involved two cycles: the first from March to April 2023 and the second from May to June 2023. Convenience sampling was used to select a sample size of 256 patients for the first cycle and 238 patients for the second cycle. Data collection involved recording patient demographics, registration and consultation times, triage categories assigned by the triage nurse, admission decisions, and independent assessment of triage accuracy by a pair of doctors.

After completing the first cycle, an educational intervention was conducted with the triage nurses, providing detailed explanations on accurate usage of the MTS and instructing them to refer non-urgent cases to the outpatient department or the Casualty Medical Officer. Circulars containing instructions regarding MTS usage were also distributed. The second cycle was then conducted, following the same data collection procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented to the Emergency Department (ED) of Medical Unit I, Benazir Bhutto Hospital, Rawalpindi.
* Patients whose data was recorded and available for analysis.
* Patients of all age groups and genders.
* Patients who visited the ED during the specified audit cycles.

Exclusion Criteria:

* Children (age<13 years)
* Patients whose data was incomplete or missing crucial information for analysis.
* Patients who were not seen by a doctor and did not receive a discharge diagnosis.
* Patients who visited the ED outside the specified audit cycles.
* Patients who were transferred to another facility before receiving triage or medical assessment.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population in this clinical audit consisted of patients who presented to the Emergency Department (ED) of Medical Unit I, Benazir Bhutto Hospital, Rawalpindi The study population encompassed patients of all age groups and genders who visited the ED during the specified audit cycles and met the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
The number of patients categorized into each triage category by the Triage Nurse | 3 months
  The study aimed to assess how effectively the triage nurses in the Emergency Department (ED) of Benazir Bhutto Hospital, Rawalpindi, categorized patients into different triage categories based on their presenting symptoms. The triage decisions made by the triage nurses were compared with the triage decisions made by the emergency physicians, using the discharge diagnosis as a benchmark. The accuracy of triage was determined by evaluating whether the assigned triage category matched the severity of the patients' condition as indicated by the discharge diagnosis. The study focused on identifying cases of under-triage, over-triage, accurate triage, and un-triage to assess the overall effectiveness of the triage process and to identify areas for improvement.
The number of patients categorized into each triage category by the ER Physician | 3 months
  The patients were categorized into triage categories by the ER Physician upon arrival to doctor (after triage from Triage counter, by the Triage Nurse). This triage was based on the discharge diagnosis and the ER Physician's evaluation.

SECONDARY OUTCOMES:
Number of patients who presented to the ER with cases that didn't require emergency management | 3 months
  A significant portion of the study focused on non-urgent cases that presented to the Emergency Department (ED). These non-urgent cases refer to patients whose medical conditions or symptoms did not require immediate or urgent medical attention. They were evaluated by two independent ER Physicians and labelled 'non-urgent' if they booth sufficiently believed this case required no emergency care and there was no jurgency to get checked by a doctor for the patient. Instead, these cases could have been appropriately managed in the outpatient setting, such as through scheduled appointments in clinics or primary care facilities
Time between patient's arrival to ER and being attended to by the doctor (waiting time) for each triage category | 3 months
  The waiting time each patient spent before they were attended to by the doctor was measured and recorded according to the triage category they belonged to.

CONTACTS AND LOCATIONS:
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD